CLINICAL TRIAL: NCT03341923
Title: Clinical Evaluation of DAILIES TOTAL 1® Multifocal Compared to 1-Day Acuvue® Moist® Multifocal in a Japanese Population
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: CLJ369-P001
Record Dates: First submitted 2017-11-09; First posted 2017-11-14 (Actual); Results first posted 2019-04-16 (Actual); Last update posted 2019-04-16 (Actual); Status verified 2019-03

CONDITIONS: Refractive Error; Presbyopia
Keywords: contact lenses; lens centration; multifocal
MeSH Terms: conditions — Refractive Errors; Presbyopia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- DT1MF, then AMMF (Other): Delefilcon A multifocal contact lenses, followed by etafilcon A multifocal contact lenses. Each product worn in both eyes for 14 +/- 3 days.
  Interventions: Device: Delefilcon A multifocal contact lenses; Device: Etafilcon A multifocal contact lenses
- AMMF, then DT1MF (Other): Etafilcon A multifocal contact lenses, followed by delefilcon A multifocal contact lenses. Each product worn in both eyes for 14 +/- 3 days.
  Interventions: Device: Delefilcon A multifocal contact lenses; Device: Etafilcon A multifocal contact lenses

INTERVENTIONS:
Device: Delefilcon A multifocal contact lenses — Silicone hydrogel multifocal contact lenses for daily disposable wear
  Other Names: DAILIES TOTAL 1® Multifocal
Device: Etafilcon A multifocal contact lenses — Hydrogel multifocal contact lenses for daily disposable wear
  Other Names: 1-DAY ACUVUE® Moist® Multifocal

SUMMARY:
The purpose of this clinical study is to evaluate DAILIES TOTAL1® Multifocal (DT1MF) contact lenses compared to 1-DAY ACUVUE® Moist® Multifocal (AMMF) contact lenses for investigator-graded lens centration in a Japanese population.

DETAILED DESCRIPTION:
Subjects will be randomly assigned to one of two sequences of investigational product wear ((DT1MF→AMMF, AMMF→DT1MF). Each product will be worn in both eyes for at least 11 days.

ELIGIBILITY:
Inclusion Criteria:

* Sign informed consent
* Habitually wear multifocal soft/ silicone hydrogel contact lenses
* Require a near spectacle ADD of +0.50 diopters (D) to +2.50D (inclusive)
* Correctable to 20/30 Snellen or 0.2 logarithm minimum angle of resolution (logMAR) or better in each eye at distance
* Willing to wear contact lenses and attend all study visits

Exclusion Criteria:

* Currently wearing DAILIES TOTAL 1® Multifocal or 1-DAY ACUVUE® Moist® Multifocal contact lenses
* Any eye condition that would make contact lens wear unadvisable
* Any use of medication that would make contact lens wear unadvisable
* Prior refractive surgery

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 151 (Actual)
Dates: Start 2017-12-20 (Actual); Primary Completion 2018-06-05 (Actual); Study Completion 2018-06-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- Japan (4):
  - Alcon Investigative Site, Koto-Ku, Tokyo
  - Alcon Investigative Site, Nakano-ku, Tokyo
  - Alcon Investigative Site, Shinagawa-Ku, Tokyo
  - Alcon Investigative Site, Taitō City, Tokyo

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from 4 study sites located in Japan.
Pre-assignment Details: Of the 151 enrolled, 17 subjects were exited as screen failures prior to randomization. This reporting group includes all randomized subjects (134).
Period: Period 1, First 14 Days of Wear
Arm/Group | DT1MF, Then AMMF | AMMF, Then DT1MF
Started | 67 | 67
Completed | 67 | 67
Not Completed | 0 | 0
Period: Period 2, Second 14 Days of Wear
Arm/Group | DT1MF, Then AMMF | AMMF, Then DT1MF
Started | 67 | 66 (Subject completed Period 1 but was discontinued before starting Period 2.)
Completed | 67 | 65
Not Completed | 0 | 1
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Population: This analysis population includes all subjects who used the investigational medical devices and provided data after the use. The lenses used at Visit 1 (baseline) for the selection of parameters are not regarded as investigational medical devices (Full Analysis Set).
Groups:
- Overall: Delefilcon A multifocal contact lenses and etafilcon A multifocal contact lenses worn during Period 1 and Period 2 in a crossover assignment, as randomized.
Arm/Group | Overall
Number analyzed (Participants) | 134
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.1 (5.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 103
  Male | 31
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Japanese | 134

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects With Investigator-graded Lens Centration of "Optimal"
Description: Lens centration was assessed by slit-lamp microscopy and graded on a 5-point scale, where 0=Optimal/Centered and 4=Severe decentration (with corneal exposure). One target eye was randomly selected for analysis.
Time Frame: Day 14, each product
Population: Full Analysis Set with data available
Measure: Number; unit: percentage of subjects
Groups:
- DT1MF: Delefilcon A multifocal contact lenses worn binocularly during Period 1 or Period 2 for 14 +/- 3 days, as randomized.
- AMMF: Etafilcon A multifocal contact lenses worn binocularly during Period 1 or Period 2 for 14 +/- 3 days, as randomized.
Arm/Group | DT1MF | AMMF
Number analyzed (Participants) | 132 | 133
percentage of subjects | 97.0 | 91.0
Statistical Analysis 1: Comparison: DT1MF vs AMMF; Test type: Non-Inferiority — Difference (DT1MF-AMMF) of percentage of subjects rated as "Optimal" was provided with two-sided 95% confidence interval (CI). If lower limit of CI was above -10% as non-inferiority criteria, non-inferiority was to be demonstrated; p = 0.0455, McNemar; Difference in proportion = 6.1, 95% CI 2-sided [0.2 to 11.9]
Statistical Analysis 2: Comparison: DT1MF vs AMMF; Test type: Superiority — After demonstrating noninferiority, if lower limit of CI was above 0% as superiority criteria, superiority was to be demonstrated; p = 0.0455, McNemar; Difference in proportion = 6.1, 95% CI 2-sided [0.2 to 11.9]

ADVERSE EVENTS:
Time Frame: Baseline through study completion, an average of 28 days
Description: Safety was assessed at each visit. This analysis population includes all data of subjects who used the investigational medical devices. Lenses used at Visit 1 (baseline) for the selection of parameters are not regarded as investigational medical devices (Safety Analysis Set, based on treatment-specific exposure). "At Risk" population for ocular Adverse Events is included with unit of "eyes."
Groups:
- DT1MF Ocular: Eyes exposed to delefilcon A multifocal contact lenses
- DT1MF Systemic: Subjects exposed to delefilcon A multifocal contact lenses
- AMMF Ocular: Eyes exposed to etafilcon A multifocal contact lenses
- AMMF Systemic: Subjects exposed to etafilcon A multifocal contact lenses
Arm/Group | DT1MF Ocular | DT1MF Systemic | AMMF Ocular | AMMF Systemic
All-Cause Mortality (participants affected / at risk) | 0/266 | 0/133 | 0/268 | 0/134
Serious Adverse Events (participants affected / at risk) | 0/266 | 0/133 | 0/268 | 0/134
Other Adverse Events (participants affected / at risk) | 88/266 | 0/133 | 82/268 | 0/134
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | DT1MF Ocular (N=266) | DT1MF Systemic (N=133) | AMMF Ocular (N=268) | AMMF Systemic (N=134)
Visual impairment (Eye disorders) | 82 | 0 | 70 | 0
Asthenopia (Eye disorders) | 24 | 0 | 14 | 0
Dry eye (Eye disorders) | 6 | 0 | 24 | 0
Ocular discomfort (Eye disorders) | 6 | 0 | 20 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.

DOCUMENTS (2):
  • Study Protocol (2018-01-22): https://cdn.clinicaltrials.gov/large-docs/23/NCT03341923/Prot_000.pdf
  • Statistical Analysis Plan (2015-03-16): https://cdn.clinicaltrials.gov/large-docs/23/NCT03341923/SAP_001.pdf